CLINICAL TRIAL: NCT03682406
Title: Pilot Study of the Collaborative Assessment and Management of Suicidality - Group (CAMS-G)
Brief Title: CAMS-G Group Therapy for Suicidal Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisville VA Medical Center (U.S. Federal Agency)
Collaborators: Rocky Mountain MIRECC for Suicide Prevention (Unknown)
Responsible Party: Principal Investigator, Lora Johnson, Research Facilitator, Louisville VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00467
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Suicide and Self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in even numbers to CAMS-G or care as usual.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will remain blinded to the treatment condition for all participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAMS-G (Experimental): CAMS-G is an group-based adaptation of the Collaborative Assessment and Management of Suicidality (CAMS) that has been developed to address perceived burdensomeness and thwarted belongingness, two drivers of suicide risk. Ongoing assessment and treatment planning are completed using the CAMS Suicide Status Form in the group modality, with involvement from group members and group facilitators. Driver-focused intervention strategies and group process also occur in the group based upon the unique needs of the group members. Groups are 90-minutes in length and occur on a weekly basis.
  Interventions: Behavioral: CAMS-G
- Care as Usual (Other): Care as usual includes access to all existing forms of treatment that currently exist at the Robley Rex VAMC and affiliated CBOCs, such as individual and group psychotherapy, suicide prevention programming and case management, psychiatric care, social work services, and substance use disorder counseling. We will essentially track the control condition over time as they engage in the typical services provided to suicidal Veterans through the Robley Rex VAMC. The CAMS-G study participants will have access to the same services delivered as part of care as usual, with the only difference being their participation in the CAMS-G treatment for suicidality.
  Interventions: Behavioral: CAMS-G

INTERVENTIONS:
Behavioral: CAMS-G — Group-based suicide-specific intervention based upon the Collaborative Assessment and Management of Suicidality.

SUMMARY:
The primary aim of this pilot study is to determine the feasibility and acceptability of CAMS-G. Our aim is to determine if CAMS-G is an effective treatment and whether it has the potential to be tested in a large-scale setting.

DETAILED DESCRIPTION:
A total of 60 patients from either the Robley Rex VAMC inpatient psychiatry unit or outpatient clinics will be enrolled in the study. If the Veteran is referred from inpatient psychiatry, study staff will meet with the Veteran to determine eligibility and consent the Veterans on the inpatient unit prior to discharge. A phone interview will be scheduled to complete the baseline interview after the Veteran has been discharged from the inpatient psychiatry unit. Outpatient referrals will be handled similarly. Whenever possible, to reduce participant burden, the study team will meet Veterans at a community based outpatient clinic (CBOC) to consent outpatients either immediately prior to or after a scheduled appointment. A phone interview will be scheduled to complete the baseline prior to the start of their group. Patients will then be randomized to either (a) an experimental group receiving CAMS-G or (b) a group receiving care as usual. All study participants will then complete telephone follow-up assessments at 1-, 3-, and 6-month time points administered by members of the research team. Dr. Gutierrez and his study team will rate the CAMS-G sessions for adherence to the treatment manual. Individual Veterans remain in the CAMS-G sessions until their suicidal crisis is resolved. The baseline assessment battery will take approximately 60 minutes and the 1-, 3-, and 6-month assessment batteries will take approximately 45 minutes.

The Client Satisfaction Questionnaire will be administered at three- and six-month follow-up for each study participant. This will allow reflection on the acceptability and perceived utility of CAMS-G. Notes will be kept on patients who decided to drop out of the intervention and/or the study. The outcome of this aim is evidence that the final CAMS-G manual and study procedures that would be used in an efficacy trial are acceptable to participants. The investigators will examine the mean and standard deviation for the total score and individual items to determine if study participants report acceptable ratings of satisfaction. The investigators will review the responses to open ended questions regarding what Veterans perceived as being helpful about their group experience and what they could do in the future if they become suicidal.

The investigators will tabulate average scores and standard deviations for the overall rating and each individual item on the CAMS-G Rating Scale to determine whether the facilitators maintained fidelity to the treatment manual over the course of the study.

The investigators will tally the different services received by study participants in order to accurately describe what care as usual consisted of for all study participants, regardless of their assigned treatment condition. This will also the investigators to control for any major differences in care as usual between treatment conditions, for example more individual psychotherapy for one condition, when examining between group differences on outcomes of interest.

At the termination of data collection, the investigators will complete a data cleansing process. Descriptive statistics for demographic and clinical variables will be tabulated. All scales will be scored and subscales described. This process will include examining the data for missing values, appropriate ranges, and outliers, with transformations to skewed data applied as needed. Although the randomization design should ensure balance between the two groups, it is essential to control for any known confounders in the design and analysis to prevent a biased assessment of the suicide assessment effect. Any baseline demographic or clinical variables found to be statistically significant in the analysis and significantly associated with the outcomes of interest will be included as covariates in all analytic models.

Dropouts and missing data. The investigators will use an intent-to-treat sample to complete our analyses. That is, all participants who provide consent, are randomized to a treatment condition, and attend at least one group therapy session will be included in the analyses regardless of whether they drop out or complete a full course of group therapy. To understand whether treatment drops were completely random, random, or informative, the investigators will analyze our missing data and adjust our interpretation of the results accordingly. The investigators will use generalized linear mixed models (GLMM) to measure differences at 1-, 3-, and 6-months follow-up between veterans in the CAMS-G treatment condition and those in the control treatment condition on constructs of Hopelessness, Thwarted Belongingness, Perceived Burdensomeness, Overall Symptom Distress, and Reasons for Living. The investigators will use Poisson or similar variant of generlized linear mixed modeling (GLMM) for skewed and count data to measure differences at 1-, 3-, and 6-months follow-up between Veterans in the CAMS-G treatment condition and those in the control treatment condition on severity of suicidal ideation and incidence of self-directed violence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18-89 years old
2. Endorses suicidality (acknowledges recent/current suicidal thoughts, plans, and/or behavior and wish to work on it clinically).
3. Veteran is willing to engage in treatment around the suicidality.
4. Eligible to receive care at the Robley Rex VA Medical Center
5. English speaking based on the need to participate in group treatment

Exclusion Criteria:

1. CAMS-G is designed to be as broadly inclusive as possible. On a case-by-case basis, psychopathology and/or cognitive limitations that significantly interfere with the patient's ability to interact effectively and/or benefit from a group intervention could preclude the patient from participating in the group.
2. A Veteran could be excluded if he or she has a circumstance that could be harmful to other members who are already in the group (e.g., we will not enroll a sex offender who is working on that issue into a group with a victim of sexual abuse).
3. A Veteran who is unwilling to meaningfully engage in treatment (e.g., unwilling to reduce access to lethal means, directly address suicidal drivers, engage in collaborative treatment planning, develop a safety plan, participate in group discussion, etc.) is inappropriate for participation in the group on an outpatient basis.
4. Veterans will be excluded if they have previously been in a CAMS-G treatment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Self-Harm Behavior Questionnaire | 6 months
  Self-report measure composed of four sections, each assessing different facets of suicidality. Each subsection will be scored for occurrence and severity, including non-suicidal self-injury, suicide attempts, suicide threats, and suicidal ideation.
Changes Beck Scale for Suicidal Ideation | 6 months
  19-item assessment used to evaluate the current intensity of the patient's specific attitudes toward, behavior, and plans to commit suicide. Total score will be reported which ranges from 0 (no suicidal ideation) to 38 (high suicidal ideation)
Changes in Interpersonal Needs Questionnaire, which measures constructs of thwarted belongingness and perceived burdensomeness | 6 months
  12-item measure of the extent to which individuals feel connected to others (i.e., belongingness) and like a burden on people in their lives (i.e., perceived burdensomeness). Subscale total scores for thwarted belongingness and perceived burdensomeness will be reported. For thwarted belongingness, scores range from 9 (low) to 63 (high). For perceived burdensomeness, scores range from 6 (low) to 42 (high).
Changes in Beck Hopelessness Scale | 6 months
  20-item true-false self-report scale that measures the level of negative expectations about the future held by respondents over the previous week. Scores range from 0 to 20 representing nil (0-3), mild (4-8), moderate (9-14), and severe (> 14) levels of hopelessness.
Changes in Reasons for Living Inventory | 6 months
  48-item measure that rates the importance of different reasons why people choose not to kill themselves. Total score will be reported, which ranges from 48 (low reasons for living) to 288 (High reasons for living).
Changes in Outcome Questionnaire-45 | 6 months
  45-item tracking/assessment instrument measuring overall symptom distress, which ranges from 0 (low distress) to 180 (high distress)
Changes in Optimism and Hope Scale | 6 months
  14-item self-report measure combining a measure of dispositional optimism and trait hopefulness, with scores ranging from 0 (low) to 42 (high)

OTHER OUTCOMES:
Group Cohesion Scale | 3 months
  9-item scale used in this study to assess participants' perceptions of how well the group members form feelings of interpersonal bonds in the group, scores range from 1 (low) to 63 (high)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lederer, MD, Study Chair — Louisville VAMC
Locations (1):
- Robley Rex VAMC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gutierrez PM, Johnson L, Podlogar MC, Hagman S, Muehler TA, Hanson J, Pierson JT, Brown AA, O'Connor S. Pilot study of the Collaborative Assessment and Management of Suicidality-Group. Suicide Life Threat Behav. 2022 Apr;52(2):244-255. doi: 10.1111/sltb.12817. Epub 2021 Nov 15. PMID 34780099